CLINICAL TRIAL: NCT04446624
Title: Analisi Dei Marcatori di Stress Ossidativo in Pazienti Affetti da Tumore Della Mammella, Sottoposte a Radioterapia Postoperatoria e Psicoterapia Con Elementi di Musicoterapia
Brief Title: Oxidative Stress, Anxiety and Depression in Breast Cancer Patients: Impact of Music Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Marco Krengli, Full Professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE 193/17
Record Dates: First submitted 2020-06-05; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Depression, Anxiety; Oxidative Stress
Keywords: Oxidative stress; Radiotherapy; Music therapy; Quality of life; Resilience; Breast cancer; Depression and anxiety
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (No Intervention): Patients in the TAU group will receive the treatment routinely offered to patients undergoing RT for breast cancer.
- Music therapy intervention (PSY) (Experimental): Patients in the PSY group will participate to a short-term group psychotherapy with elements of music therapy; meetings will be 1 / week, for a total of 6 weeks. Beginning of psychotherapy intervention will be 1-2 weeks after recruitment at T0 and will therefore cover the entire duration of the RT cycle.
  Interventions: Other: Music therapy intervention

INTERVENTIONS:
Other: Music therapy intervention — Group psychotherapy with music intervention
  Arms: Music therapy intervention (PSY)

SUMMARY:
Oxidative stress plays an important role in the development of breast cancer, and also of depression which can affect the ability to deal with cancer.

The main objective of this study is to evaluate the impact of a group psychotherapy with elements of music therapy in a population of patients suffering from breast cancer, treated with surgery and undergoing post-operative RT.

Study outcomes will be the following:

1. Effectiveness of the proposed intervention especially on anxiety and depression, as described by changes in psychometric test scores.
2. Changes of oxidative stress and inflammation markers, such as high sensitivity C-reactive protein (hs-PCR), fibrinogen and lipoprotein-associated phospholipase A2 (Lp-LPLA2), GSH, TBARS, IL4, IL6, TNF-α, α and γ tocopherol, carotenoids, folic acid, vitamin B12.
3. Correlation between changes of markers (see point 2) and the clinical/psychometric variables under study.

Methods This is a prospective randomized monocentric study, which will involve patients diagnosed with early stage invasive breast cancer (pTis-1-2 N0-1 M0), who underwent conservative surgery, and candidates for adjuvant RT. Patients will be identified during the RT visit. Patients who meet the eligibility criteria and who have signed informed consent will be randomized (1:1) as follows: group supportive psychotherapy with elements of music therapy (PSY); control group - treatment as usual (TAU ). Patients will undergo psychometric assessment and blood sampling (10 ml) at T0 (baseline), T1 (last day of RT), T2 (3 months after the end of RT).

Study duration will be one year; during the first 9 months, patients will be recruited and treated, in the following period follow-up evaluations will be completed and data analyses will be conducted.

Sample size Based on literature data, indicating average anxiety ranges measured with a STAI score from 43.4 to 46.2 and assuming, in the experimental group, a clinically significant reduction of 9 points (Bulfone 2009, Rossetti 2017), 24 patients per group have to be enrolled (alpha: 0.05; Beta: 0.20).

Statistical analysis A simple randomization in 1:1 ratio will be carried out. Differences between the 2 groups will be used to assess the impact of psychotherapy intervention with elements of music therapy. A descriptive statistical analysis and estimate of relative risks will be performed.

DETAILED DESCRIPTION:
Background

Mood alterations, particularly depression, are defined by the National Comprehensive Cancer Network (NCCN) as "multi-factorial unpleasant emotional experiences of psychological (cognitive, behavioral, emotional), social and/or spiritual nature that may interfere with the ability to cope with cancer, its physical symptoms and treatment". A recent meta-analysis showed that 8% to 24% of cancer patients in non-palliative care settings experienced depression. Many factors may contribute to depression in breast cancer patients, including age at diagnosis, cancer stage, surgery, and chemotherapy. Inflammation and oxidative stress are considered possible causing factors for mood disorder in patients with breast cancer, who show an increase in plasma rate of TNF alpha, IL6 and NFKB; alterations in the plasma levels of antioxidant agents, such as glutathione (GSH) and vitamin C, may be found as well. Correlation between mood alterations and oxidative stress is a frequently discussed topic in the scientific literature. Oxidative stress plays a key role in breast cancer development. In patients with different stages of breast cancer it was found a direct correlation between serum total oxidant status (TOS), total antioxidant status (TAS), oxidant stress index (OSI) and cancer progression. In particular, TOS and OSI gradually increase as the disease progresses, while TAS diminishes. Lipoprotein-associated phospholipase A2 (Lp-LPLA2) plays an important role in inflammation, but also in cytokine-induced depression and sickness behavior. Lp-PLA2 could be an important link between lipid homeostasis, inflammatory vascular response and depression. Thus, the analysis of Lp-PLA2 levels associated with LDL in patients with breast cancer, never performed before in the literature, could act as an important system for assessing the inflammatory status of this population.

The potential predictive factors of depression during and after radiotherapy (RT) remains largely unexplored or analysed in retrospective studies or with limited numbers of patients. The perception of stigma could have an impact on depressive symptoms in cancer patients. More depressive symptoms, fatigue and stress and higher levels of inflammation markers may be found in patients with a history of childhood trauma. Another factor that has shown a significant association with depression is the role of post-surgical and post-RT aesthetic changes in women with breast cancer, while depressive symptoms were not influenced by RT toxicity.

To date, however, prospective studies are needed to identify primary risk factors for depression in patients with breast cancer treated with RT. A proposed mechanism linking radiation therapy and depression is inflammation. Markers of inflammation are increased in patients with depression, and blockage of inflammation mechanisms can also modulate depressive symptoms, in particular "fatigue" in cancer patients. To date only one study has evaluated this relationship, quantifying the expression of IL6 receptors in patients with depression. In general, studies confirmed an improvement in anxiety and depression with the progress of the radiant treatment, and chronic changes occurred only in a percentage of about 10% of the patients.

Oxidative stress seems to play also an important role in the aetiology of adverse effects from radiation therapy.

Mood alterations, depression in particular, negatively affect both RT, in which the patient's "compliance" plays a fundamental role, and the patient's quality of life.

The need for psychological / psychotherapeutic support in cancer patients, and in particular in breast cancer patients, is known and discussed in the literature, and there are many studies about integrative therapeutic approaches.

Among the therapeutic approaches for the treatment of depression, analytical receptive music therapy, both as individual or group therapy, has been assessed; it consists in listening to music and in the subsequent verbalization of experiences, emotions and images aroused. A group music therapy intervention has recently proved to be more effective than a control intervention in breast cancer women treated with chemotherapy.

The recent "Clinical Practice Guidelines" on the "evidence-based" use of integrative therapies during and after treatment for breast cancer has supported the use of various integrative therapy approaches. Music therapy has been recommended to reduce anxiety and stress, and also in case of depression and mood disorders. It should also be noted that in a recent study, the improvement of symptoms in a group of patients suffering from depression was accompanied by an increase in anti-inflammatory cytokines such as IL4.

Objectives The main objective is to evaluate the impact of a group psychotherapy with elements of music therapy, in a population of patients suffering from breast cancer, treated with surgery and undergoing post-operative RT.

Selection criteria Subjects Patients diagnosed with early stage invasive breast cancer (pTis-1-2 N0-1 M0), who underwent conservative surgery, and candidates for adjuvant RT. Patients will be identified during the RT visit and assessed according to inclusion and exclusion criteria, detailed elsewhere.

The study does not include modifications in the standard surgical and RT process of the healthcare facility.

At any time during the study, the patient can withdraw the consent to participate and leave the study.

During the entire study period, the patient will be treated according to the standards of Good Clinical Practice (Declaration of Helsinki).

Patients who meet the eligibility criteria and who have signed informed consent will be randomized (1:1) into 2 groups:

1. group undergoing group psychotherapy with elements of music therapy (PSY)
2. control group - treatment as usual (TAU). Timing

All enrolled patients will be assessed with psychometric assessment and blood sampling (10 ml) at Time T0 (pre-RT), Time T1 (last day of RT), Time T2 (3 months after the end of RT).

Procedures

The patients will be randomized into two groups:

treatment as usual (TAU) group psychotherapy (PSY) Specifically, patients in the TAU group will receive the treatment routinely offered to patients undergoing RT for breast cancer.

The radiation therapy treatment will be performed at the SC Radiotherapy of the AOU "Maggiore della Carità" in Novara.

The treatment consists in the irradiation of the entire residual breast volume. The irradiation technique will be established according to the current standards of the SC Radiotherapy which include a conformal 3D RT (3D-CRT) or an RT with intensity modulation (IMRT). The treatment will be performed using 6 and 15 MV photon beams produced by a linear accelerator. RT sessions will be performed daily from Monday to Friday for a total of 20-25 sessions. The current protocol provide a total prescribed dose of: 45 Gy, 2.25 Gy/die with boost dose on the neoplastic bed by sequential electron beam or concomitant photon beams or 50 Gy, 2 Gy/die.

Every five RT sessions, patients will receive a clinical evaluation by the oncologist radiotherapist.

The patients in the PSY group will participate to a short-term group psychotherapy with elements of music therapy; meetings will be 1 / week, for a total of 6 weeks. Beginning of psychotherapy intervention will be 1-2 weeks after recruitment at T0 and will therefore cover the entire duration of the RT cycle. Psychotherapy meetings will take place at the SCDU Psychiatry of the AOU Maggiore della Carità.

Obviously, according to ethical reasons, in case a patient in each group (TAU, PSY) at any time, needs a psychiatric visit, psychopharmacological support or individual support, this will be offered according to clinical indications. If these interventions are started before the completion of the protocol, the patient will continue for ethical reasons the intervention started (and in addition the intervention considered necessary by the clinician) and the planned evaluations, but she will be excluded from the analyses on the effectiveness of the proposed intervention, because of the bias of additional treatments.

Similarly, according to ethical reasons, if patients at the end of the protocol need additional psychotherapeutic and/or pharmacological support, this will be offered according to clinical conditions that could be different for each patient. This will not imply exclusion from the study protocol.

Psychiatric evaluation

Depressive symptoms - Beck Depression Inventory (BDI-II); Montgomery-Asberg Depression Rating Scale (MADRS); State-Trait Anxiety Inventory 1 and 2 (STAI Y1, STAI Y2); Resilience Scale for Adults (RSA); Short Form-36 (SF-36).

Blood samples Blood samples dosing plasma markers necessary for the study will be gathered in all patients, at the SC Radiotherapy. Samples will then be centrifuged, and serum obtained will be divided into five samples for each detection and stored at -80C, at the Physiology laboratory of the Piemonte Orientale University. The fibrinogen dosage will be included in the BCS® XP system (Siemens Healthcare Diagnostics). Dosage of α and γ of tocopherol, carotenoids, folic acid, vitamin B12 will finally be performed using high resolution liquid chromatography (Agilent 1200 Series). Measurements of the plasma glutathione rate (GSH), lipid peroxidation products (TBARS), IL4, IL6 and TNF alfa will be included in widely used kits. The measurements will be carried out at the Physiology laboratory of the Piemonte Orientale University by Biotechnologists under the supervision of Prof. Elena Grossini.

Population Sample size Based on literature data, indicating average anxiety ranges measured with a STAI score from 43.4 to 46.2 and assuming, in the experimental group, a clinically significant reduction of 9 points, 24 patients per group have to be enrolled (alpha: 0.05; Beta: 0.20). In consideration of this data, a sample of 60 total patients is assumed.

Statistical analysis A simple randomization in 1:1 ratio will be carried out through a special statistical program. Differences between the 2 groups will be used to assess the impact of the psychotherapy intervention with elements of music therapy. A descriptive statistical analysis and estimate of relative risks will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1
* Age > 18 years
* Histologically confirmed invasive / intraductal breast cancer
* Conservative breast surgery (quadrantectomy, nodulectomy)
* Free surgical margins
* Pathological stage pTis, pT1-2 pN0-1 M0 (according to the TNM classification)
* Indication for adjuvant RT
* Signature of informed consent

Exclusion Criteria:

* Age < 18 years
* indication to chemotherapy / targeted therapy
* diagnosis of previous major depressive episode
* current comorbidity with abuse of alcohol and / or psychotropic substances
* ongoing psychopharmacological treatment with antidepressants and / or mood stabilizers
* diagnosis of mental retardation, dementia, or other cognitive impairment
* autoimmune / inflammatory diseases / diabetes mellitus
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in anxiety from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  Anxiety is assessed with the State-Trait Anxiety Inventory 1 and 2 (STAI Y1, STAI Y2), a 40-item self-administered test for the assessment of state and trait anxiety. Each item is rated 1 to 4 (1= not at all, 4= severe); no specific cut-off scores exist. The highest the score, the greater is anxiety.
Change in depression from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  Depression is assessed with the Montgomery-Asberg Depression Rating Scale (MADRS and with the Beck Depression Inventory (BDI). The MADRS is a 10-item clinician-rated scale for depressive symptoms detection and severity assessment. Each item is rated on a six-point scale, hence 60 is the maximum total score indicating the maximum severity of depressive symptoms. A score <6 points stands for no depression (normal), 7-19 mild depression, 20-34 moderate depression, ≥ 35 severe depression. The BDI is a 21-item self-administered test for the evaluation of subjective depressive feelings or symptoms. It is rated on a 4-points scale (from 0 to 3 according to severity), with the following cutoff values: 0-9 minimal depression, 10-18 mild depression, 19-29 moderate depression, 30-63 severe depression.
Change in Glutathione (GSH) from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  GSH measurement was performed through the Glutathione Assay Kit (Cayman Chemical, Ann Arbor, MI, USA). For the experiments, each plasma sample was deproteinated and centrifuged at 2000 g for 2 min. Fifty μl of the samples was transferred to a 96-well plate where GSH was detected through a spectrophotometer (VICTOR™ X Multilabel Plate Reader), at excitation/emission wavelengths of 405-414 nm. To ensure accurate GSH quantification (expressed as µM), a reference curve with the GSH Standard was prepared (range of known GSH concentration: 0-16 μM). As regards the performance of the assay, variation coefficient of 3.6% for inter-assay and 1.6% for intra-assay is reported.
Change in TBARS from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  TBARS were determined as malonyldialdeide (MDA) release. MDA measurement was performed by using the TBARS assay Kit (Cayman Chemical). For the experiments, 100 µl of each plasma sample was added to 100 µl of sodium dodecyl sulfate (SDS) solution and 2 ml of the Color Reagent. After centrifugation, 150 μl of each sample was transferred to a 96-well plate where MDA was detected through a spectrophotometer (VICTOR™ X Multilabel Plate Reader), at excitation/emission wavelengths of 530-540 nm. In order to quantify the correct values of TBARS (expressed as µM MDA), a reference standard curve was prepared (range of known TBARS concentration: 0-50 μM). As regards the performance of the assay, intra-coefficient of variation of 5.5% and an inter-coefficient variation of 5.9% is reported.

SECONDARY OUTCOMES:
Change in resilience from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  Resilience is assessed with the Resilience Scale for Adults (RSA). This is a 33-item self-administered scale evaluating intra- or inter-relational stress preventing factors (positive self-perception, positive future perception, social competence, structured style, family cohesion and social resources). The higher is the total score, the greater is the subject's resilience.
Change in quality of life from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  Quality of life is assessed with the Short Form-36 (SF-36), a self-administered test assessing health-related quality of life, both from a somatic and psychological standpoint. It assesses several sub-areas: physical activity, role and physical health, physical pain, general health, vitality, social activities, role and emotional state, mental health and health change. Results are expressed in age- calculated percentiles.
Change in Human IL-6 from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  IL-6 measurement was performed by using the Human IL-6 ELISA kit (Invitrogen Carlsbad, California, USA). For the experiments, 50 μl of each plasma sample and 50 μl of Assay Buffer 1X were added to each well, with 50 μl of Biotin-Conjugate and incubated at room temperature (RT) on microplate shaker for 2 h. After addition of 400 μl Wash Buffer, 100 μl Streptavidin-HRP and 100 μl Substrate Solution, each well was incubated for 10 min at RT in the dark. The enzyme reaction was stopped by adding 100 μl Stop Solution, and IL-6 was detected through a spectrophotometer (VICTOR™ X Multilabel Plate Reader), using a wavelength of 450 nm. In order to quantify the correct value of IL-6 in each sample (expressed as pg/ml), a reference standard curve was prepared (range of IL-6 standard concentration:0-20 pg/mL). As regards the performance of the assay, intra-coefficient of variation of 8.5% and an inter-coefficient variation of 9.8% is reported. The sensitivity of the test is < 1 pg/ml.
Change in Human TNFα from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  TNFα measurement was performed with the Human TNF alpha ELISA kit (Invitrogen, Carlsbad, California, USA). For the experiments, 50 μl of each plasma sample and 50 μl of Sample Diluent were added to each well, with 50 μl of Biotin-Conjugate and incubated at RT on microplate shaker for 2 h. After addition of 400 μl Wash Buffer, 100 μl Streptavidin-HRP and 100 μl Substrate Solution, each well was incubated for 10 min at RT in the dark. The enzyme reaction was stopped by adding 100 μl of Stop Solution and each well was read immediately. TNFα was detected through a spectrophotometer (VICTOR™ X Multilabel Plate Reader), using a wavelength of 620 nm. To quantify the correct value of in each sample, a reference standard curve was prepared (range of TNFα standard concentration: 0-100 pg/mL). As regards the performance of the assay, intra-coefficient of variation of 3.4% and inter-coefficient variation of 5.2% is reported. The sensitivity of the test is 0.13 pg/ml.
Change in Retinol, α and γ -tocopherol, lycopene and β carotene from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  HPLC analysis of retinol, α and γ -tocopherol, lycopene and β carotene were carried out on Agilent 1200 series HPLC.
  200 ml of each plasma sample was mixed with 300µl of water and 500 µl of ice-cold absolute ethanol and immediately vortexed for 10 s. Two millilitres of ice-cold hexane was added. The mixture was immediately vortexed for 2 minutes and then centrifuged at 3000 g for 1 min and 1 ml of the upper (organic) layer was transferred in a vial, evaporated to dryness under a nitrogen stream and reconstituted with 100 ml of a mixture of acetonitrile/dichloromethane/methanol for HPLC analysis.
  Twenty microlitres of this mixture were then injected and the antioxidants were eluted with a mobile phase containing acetonitrile/dichloromethane/methanol, glacial acetic acid (1 g /l) at a constant flow of 1.8 ml/min.
  Detection of lipid soluble antioxidants was performed at specific wavelength: retinol (326 nm), γ- and α-tocopherol (292nm), lycopene and β-carotene (460nm).
Change in Cholesterol and high sensitivity C-reactive Protein from baseline to follow-up | Time T0 (pre-RT); Time T1 (through RT completion, an average of 27 days); Time T2 (3 months after the end of RT)
  Colesterol and high sensitivity C-reactive Protein (CRP) were analyzed on ADVIA® 1800 Clinical Chemistry Analyzer (Siemens Healthcare Diagnostics), by automated methods and certified kits.
  Colesterol (range:0 - 200 mg/dL) High sensitivity C-reactive Protein (range:0 - 1 mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Krengli, MD, Study Chair — University of Piemonte Orientale
Locations (1):
- Department of Translational Medicine, Università del Piemonte Orientale, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Bidstrup PE, Christensen J, Mertz BG, Rottmann N, Dalton SO, Johansen C. Trajectories of distress, anxiety, and depression among women with breast cancer: Looking beyond the mean. Acta Oncol. 2015 May;54(5):789-96. doi: 10.3109/0284186X.2014.1002571. Epub 2015 Mar 11. PMID 25761086
- [Background] Bower JE. Behavioral symptoms in patients with breast cancer and survivors. J Clin Oncol. 2008 Feb 10;26(5):768-77. doi: 10.1200/JCO.2007.14.3248. PMID 18258985
- [Background] Brunault P, Suzanne I, Trzepidur-Edom M, Garaud P, Calais G, Toledano A, Camus V. Depression is associated with some patient-perceived cosmetic changes, but not with radiotherapy-induced late toxicity, in long-term breast cancer survivors. Psychooncology. 2013 Mar;22(3):590-7. doi: 10.1002/pon.3038. Epub 2012 Feb 7. PMID 22315168
- [Background] Bulfone T, Quattrin R, Zanotti R, Regattin L, Brusaferro S. Effectiveness of music therapy for anxiety reduction in women with breast cancer in chemotherapy treatment. Holist Nurs Pract. 2009 Jul-Aug;23(4):238-42. doi: 10.1097/HNP.0b013e3181aeceee. PMID 19574761
- [Background] Carr CE, O'Kelly J, Sandford S, Priebe S. Feasibility and acceptability of group music therapy vs wait-list control for treatment of patients with long-term depression (the SYNCHRONY trial): study protocol for a randomised controlled trial. Trials. 2017 Mar 29;18(1):149. doi: 10.1186/s13063-017-1893-8. PMID 28356125
- [Background] Chen SC, Chou CC, Chang HJ, Lin MF. Comparison of group vs self-directed music interventions to reduce chemotherapy-related distress and cognitive appraisal: an exploratory study. Support Care Cancer. 2018 Feb;26(2):461-469. doi: 10.1007/s00520-017-3850-1. Epub 2017 Aug 10. PMID 28799076
- [Background] Deantonio L, Cozzi S, Tunesi S, Brambilla M, Masini L, Pisani C, Gambaro G, Magnani C, Krengli M. Hypofractionated radiation therapy for breast cancer: long-term results in a series of 85 patients. Tumori. 2016 Aug 3;102(4):398-403. doi: 10.5301/tj.5000511. Epub 2016 May 26. PMID 27230276
- [Background] Esser P, Mehnert A, Johansen C, Hornemann B, Dietz A, Ernst J. Body image mediates the effect of cancer-related stigmatization on depression: A new target for intervention. Psychooncology. 2018 Jan;27(1):193-198. doi: 10.1002/pon.4494. Epub 2017 Aug 1. PMID 28685499
- [Background] Faller H, Brahler E, Harter M, Keller M, Schulz H, Wegscheider K, Weis J, Boehncke A, Reuter K, Richard M, Sehner S, Koch U, Mehnert A. Unmet needs for information and psychosocial support in relation to quality of life and emotional distress: A comparison between gynecological and breast cancer patients. Patient Educ Couns. 2017 Oct;100(10):1934-1942. doi: 10.1016/j.pec.2017.05.031. Epub 2017 May 24. PMID 28592366
- [Background] Fancourt D, Perkins R, Ascenso S, Carvalho LA, Steptoe A, Williamon A. Effects of Group Drumming Interventions on Anxiety, Depression, Social Resilience and Inflammatory Immune Response among Mental Health Service Users. PLoS One. 2016 Mar 14;11(3):e0151136. doi: 10.1371/journal.pone.0151136. eCollection 2016. PMID 26974430
- [Background] Feng JF, Lu L, Dai CM, Wang D, Yang YH, Yang YW, Liu YS. Analysis of the diagnostic efficiency of serum oxidative stress parameters in patients with breast cancer at various clinical stages. Clin Biochem. 2016 Jun;49(9):692-698. doi: 10.1016/j.clinbiochem.2016.02.005. Epub 2016 Feb 18. PMID 26899366
- [Background] Friborg O, Hjemdal O, Rosenvinge JH, Martinussen M. A new rating scale for adult resilience: what are the central protective resources behind healthy adjustment? Int J Methods Psychiatr Res. 2003;12(2):65-76. doi: 10.1002/mpr.143. PMID 12830300
- [Background] Furmaniak AC, Menig M, Markes MH. Exercise for women receiving adjuvant therapy for breast cancer. Cochrane Database Syst Rev. 2016 Sep 21;9(9):CD005001. doi: 10.1002/14651858.CD005001.pub3. PMID 27650122
- [Background] Greenlee H, DuPont-Reyes MJ, Balneaves LG, Carlson LE, Cohen MR, Deng G, Johnson JA, Mumber M, Seely D, Zick SM, Boyce LM, Tripathy D. Clinical practice guidelines on the evidence-based use of integrative therapies during and after breast cancer treatment. CA Cancer J Clin. 2017 May 6;67(3):194-232. doi: 10.3322/caac.21397. Epub 2017 Apr 24. PMID 28436999
- [Background] Han TJ, Felger JC, Lee A, Mister D, Miller AH, Torres MA. Association of childhood trauma with fatigue, depression, stress, and inflammation in breast cancer patients undergoing radiotherapy. Psychooncology. 2016 Feb;25(2):187-93. doi: 10.1002/pon.3831. Epub 2015 May 14. PMID 25976322
- [Background] Krebber AM, Buffart LM, Kleijn G, Riepma IC, de Bree R, Leemans CR, Becker A, Brug J, van Straten A, Cuijpers P, Verdonck-de Leeuw IM. Prevalence of depression in cancer patients: a meta-analysis of diagnostic interviews and self-report instruments. Psychooncology. 2014 Feb;23(2):121-30. doi: 10.1002/pon.3409. Epub 2013 Sep 16. PMID 24105788
- [Background] Lewis F, Merckaert I, Lienard A, Libert Y, Etienne AM, Reynaert C, Slachmuylder JL, Scalliet P, Paul VH, Coucke P, Salamon E, Razavi D. Anxiety and its time courses during radiotherapy for non-metastatic breast cancer: a longitudinal study. Radiother Oncol. 2014 May;111(2):276-80. doi: 10.1016/j.radonc.2014.03.016. Epub 2014 Apr 17. PMID 24746573
- [Background] Lindqvist D, Dhabhar FS, James SJ, Hough CM, Jain FA, Bersani FS, Reus VI, Verhoeven JE, Epel ES, Mahan L, Rosser R, Wolkowitz OM, Mellon SH. Oxidative stress, inflammation and treatment response in major depression. Psychoneuroendocrinology. 2017 Feb;76:197-205. doi: 10.1016/j.psyneuen.2016.11.031. Epub 2016 Nov 30. PMID 27960139
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Moreira EG, Correia DG, Bonifacio KL, Moraes JB, Cavicchioli FL, Nunes CS, Nunes SOV, Vargas HO, Barbosa DS, Maes M. Lowered PON1 activities are strongly associated with depression and bipolar disorder, recurrence of (hypo)mania and depression, increased disability and lowered quality of life. World J Biol Psychiatry. 2019 Jun;20(5):368-380. doi: 10.1080/15622975.2017.1322219. Epub 2017 May 30. PMID 28441923
- [Background] Oglodek EA. Evaluation of ADMA, carbonyl groups, CAT and NKA in depressed patients with and without posttraumatic stress disorder. Pharmacol Rep. 2017 Aug;69(4):730-737. doi: 10.1016/j.pharep.2017.02.015. Epub 2017 Feb 20. PMID 28554099
- [Background] Pariante CM. Why are depressed patients inflamed? A reflection on 20 years of research on depression, glucocorticoid resistance and inflammation. Eur Neuropsychopharmacol. 2017 Jun;27(6):554-559. doi: 10.1016/j.euroneuro.2017.04.001. Epub 2017 May 4. PMID 28479211
- [Background] Raglio A. [The efficacy of music and music therapy in the neuromotor rehabilitation]. G Ital Med Lav Ergon. 2012 Jan-Mar;34(1):85-90. Italian. PMID 22697039
- [Background] Rosenson RS, Stafforini DM. Modulation of oxidative stress, inflammation, and atherosclerosis by lipoprotein-associated phospholipase A2. J Lipid Res. 2012 Sep;53(9):1767-82. doi: 10.1194/jlr.R024190. Epub 2012 Jun 4. PMID 22665167
- [Background] Rossetti A, Chadha M, Torres BN, Lee JK, Hylton D, Loewy JV, Harrison LB. The Impact of Music Therapy on Anxiety in Cancer Patients Undergoing Simulation for Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Sep 1;99(1):103-110. doi: 10.1016/j.ijrobp.2017.05.003. Epub 2017 May 8. PMID 28816136
- [Background] Su KP, Huang SY, Peng CY, Lai HC, Huang CL, Chen YC, Aitchison KJ, Pariante CM. Phospholipase A2 and cyclooxygenase 2 genes influence the risk of interferon-alpha-induced depression by regulating polyunsaturated fatty acids levels. Biol Psychiatry. 2010 Mar 15;67(6):550-7. doi: 10.1016/j.biopsych.2009.11.005. Epub 2009 Dec 24. PMID 20034614
- [Background] Torres MA, Pace TW, Liu T, Felger JC, Mister D, Doho GH, Kohn JN, Barsevick AM, Long Q, Miller AH. Predictors of depression in breast cancer patients treated with radiation: role of prior chemotherapy and nuclear factor kappa B. Cancer. 2013 Jun 1;119(11):1951-9. doi: 10.1002/cncr.28003. Epub 2013 Mar 19. PMID 23512358
- [Background] Vollbracht C, Schneider B, Leendert V, Weiss G, Auerbach L, Beuth J. Intravenous vitamin C administration improves quality of life in breast cancer patients during chemo-/radiotherapy and aftercare: results of a retrospective, multicentre, epidemiological cohort study in Germany. In Vivo. 2011 Nov-Dec;25(6):983-90. PMID 22021693
- [Background] Wagner LI, Pugh SL, Small W Jr, Kirshner J, Sidhu K, Bury MJ, DeNittis AS, Alpert TE, Tran B, Bloom BF, Mai J, Yeh A, Sarma K, Becker M, James J, Bruner DW. Screening for depression in cancer patients receiving radiotherapy: Feasibility and identification of effective tools in the NRG Oncology RTOG 0841 trial. Cancer. 2017 Feb 1;123(3):485-493. doi: 10.1002/cncr.29969. Epub 2016 Nov 10. PMID 27861753
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Zhang M, Huang L, Feng Z, Shao L, Chen L. Effects of cognitive behavioral therapy on quality of life and stress for breast cancer survivors: a meta-analysis. Minerva Med. 2017 Feb;108(1):84-93. doi: 10.23736/S0026-4806.16.04528-6. Epub 2016 Sep 16. PMID 27635602
- [Background] Spielberger CD. Inventario per l'ansia di "stato" e di "tratto", Nuova versione italiana dello S.T.A.I.-Forma Y, Organizzazione Speciali-Firenze, (1989). doi.org/10.1002/9780470479216.corpsy0943.
- [Background] Beck AT, Steer RA, Brown GK et al. BDI-II, Beck Depression Inventory: manual. San Antonio, Texas: Psychological Corp.; Boston: Harcourt Brace, ©1996
- [Background] Gramaglia C, Gambaro E, Vecchi C, Licandro D, Raina G, Pisani C, Burgio V, Farruggio S, Rolla R, Deantonio L, Grossini E, Krengli M, Zeppegno P. Outcomes of music therapy interventions in cancer patients-A review of the literature. Crit Rev Oncol Hematol. 2019 Jun;138:241-254. doi: 10.1016/j.critrevonc.2019.04.004. Epub 2019 Apr 5. PMID 31121392